CLINICAL TRIAL: NCT01086176
Title: The Impact of Post-tetanic Count on Subsequent Train-of-four During Recovery From Rocuronium
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Louis-Philippe Fortier MD Msc, HMR
Other Study IDs: MaisonneuveRH-09092
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-03

CONDITIONS: Post-tetanic Count on One Arm, the Other Arm is the Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient-control
  Interventions: Device: NMT (a device that can do neurostimulation and can record the response on the stimulation by Datex)

INTERVENTIONS:
Device: NMT (a device that can do neurostimulation and can record the response on the stimulation by Datex) — on one side, we do a post-tetanic count, on the other side we don't, after, we do train-of-four on both sides and check the difference

SUMMARY:
The purpose of this study is to see how long does the effect of a post-tetanic facilitation last on subsequent train-of-four. The investigators hypothesis is that the effect last at least 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patient having general anesthesia in dorsal decubitus with both arm available for at least an hour and a half

Exclusion Criteria:

* Age >75 or <18
* Neuromuscular disease
* difficult laryngoscopy predicted
* Allergy to rocuronium
* Malignant hyperthermia
* Full stomach
* Drugs the influence neuromuscular blockers
* Decision of the clinician to exclude his patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Poeple having general anesthesia at HMR
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The difference at 30 minutes after the post-tetanic count between the TOF% in both arms, we expect a difference of more than 10%

SECONDARY OUTCOMES:
The difference at 30 minutes after the post-tetanic count on the T1% (of the calibrated T1) in both arms, we expect a difference of more than 10%
The difference of the slope of recuperation on TOF and T1% after a post-tetanic count vs the control arm that had no tetanic stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada